CLINICAL TRIAL: NCT01779921
Title: Treatment of Congenital Factor VII Deficiency. A Prospective Observational Study
Brief Title: Treatment of Congenital Factor VII Deficiency
Acronym: F7CONDEF
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7HAEM-3578
Record Dates: First submitted 2013-01-15; First posted 2013-01-30 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Congenital Bleeding Disorder; Congenital FVII Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma for assaying of inhibiting antibodies to FVII. All samples, which are analysed at the local hospital laboratory, are to be stored and destroyed according to local rules. Inhibitor samples analysed at the central laboratory will be stored until data validation has taken place at the end of the study after which the samples will be destroyed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FVII
  Interventions: Drug: activated recombinant human factor VII; Drug: Fresh frozen plasma (Source unspecified); Drug: Plasma-derived FVII (LFB); Drug: Prothrombin Complex conc. (PCC); Drug: Plasma-derived FVII conc. (pdFVII Baxter); Drug: Plasma-derived FVII conc. (pdFVII PFL)

INTERVENTIONS:
Drug: activated recombinant human factor VII — Treatment of bleeding episodes and treatment during surgery and prophylaxis as per discretion of the investigator.
Drug: Fresh frozen plasma (Source unspecified) — Treatment of bleeding episodes and treatment during surgery and prophylaxis as per discretion of the investigator.
Drug: Plasma-derived FVII (LFB) — Treatment of bleeding episodes and treatment during surgery and prophylaxis as per discretion of the investigator.
Drug: Prothrombin Complex conc. (PCC) — Treatment of bleeding episodes and treatment during surgery and prophylaxis as per discretion of the investigator.
Drug: Plasma-derived FVII conc. (pdFVII Baxter) — Treatment of bleeding episodes and treatment during surgery and prophylaxis as per discretion of the investigator.
Drug: Plasma-derived FVII conc. (pdFVII PFL) — Treatment of bleeding episodes and treatment during surgery and prophylaxis as per discretion of the investigator.

SUMMARY:
This study is conducted globally. The aim of this study is to describe the treatment modalities and outcomes of bleeding episodes, surgery and prophylaxis in patients with factor VII (FVII) deficiency in addition to evaluate the presence (in already treated patients) and/or the appearance of inhibiting antibodies to FVII and/or therapy-related thrombosis.

Due to a Novo Nordisk commitment to the Committee for Medicinal Products for Human Use (CHMP), Novo Nordisk receives data on treatment with activated recombinant human FVII (rFVIIa, NovoSeven®) in patients with FVII deficiency from the Seven Treatment Evaluation Registry (STER, NCT01269138). These patients can also have been treated with other haemostatics for systemic administration.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by the patient or next of kin or legally acceptable representative to collect data on treatment of a given bleeding episode, surgical event or prophylactic regimen as specified in the protocol. If informed consent is provided by the next of kin or legally acceptable representative, consent must also be obtained from the patient as soon as he/she is able to do so. Informed consent should preferentially be obtained before initiation of treatment or as a minimum before entry of data into the database
* Any patient with a FVII deficiency for whom treatment of bleeding episodes, prevention related to surgery and primary/secondary prophylaxis is considered necessary by the treating physician can be enrolled
* Patients with FVII deficiency without any immediate need for treatment will be entered as stand by registered patients with capture of baseline- and demographic data only. Admission data is entered once an event occurs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with FVII deficiency (levels of FVII less than 50% of normal or a mutation known to be associated to a FVII deficiency) can be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2005-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Treatment of bleeding episodes at clinic/hospital: Treatment efficacy evaluation for each treatment modality: excellent, effective, partly effective, ineffective, or not evaluable | Evaluated at 6 hours
Treatment of bleeding episodes at clinic/hospital: Treatment efficacy evaluation for each treatment modality: excellent, effective, partly effective, ineffective, or not evaluable | Evaluated after 30 days
Treatment of bleeding episodes at clinic/hospital: Time to achieve arrest of bleeding | Time to achieve arrest of bleeding
Treatment of bleeding episodes at clinic/hospital: Number of re-bleeding episodes | Within 5 days after first product administration
Treatment of bleeding episodes at home: Treatment efficacy evaluation for each treatment modality: excellent, effective, partly effective, ineffective, or not evaluable | Evaluated at 6 hours
Treatment of bleeding episodes at home: Time to achieve arrest of bleeding | Time to achieve arrest of bleeding
Treatment efficacy (of first and/or second treatment modality) evaluated after surgery: good, partially effective, not evaluable, or ineffective | After surgery
Treatment efficacy (of first and/or second treatment modality) evaluated after surgery: good, partially effective, not evaluable, or ineffective | Evaluated after 30 days
Estimated blood loss volume | During surgery/delivery
Number of red blood cell units administered | During surgery
Number of days spent in hospital | Until last data collection (20 Jan 2012)
Number of re-bleeding episodes (associated with the surgery) | Within 5 days after surgery
Prophylactic treatment efficacy evaluation: excellent, excellent, partially effective, or effective | 30 days after first prophylaxis dose

SECONDARY OUTCOMES:
Number of bleeding episodes during prophylaxis per year | Up to one year
Number of intensive care unit (ICU) and/or the number of ward days | After first haemostatic product administration until day 30
Mortality | Within a 30-day (follow-up) period
Changes in laboratory parameters (prothombin time/international normalized ratio, activated partial thromboplastin time, FVII clotting activity, platelet count, fibrinogen) | Prior to dosing
Changes in laboratory parameters (prothombin time/international normalized ratio, activated partial thromboplastin time, FVII clotting activity, platelet count, fibrinogen) | After 15 minutes
Changes in laboratory parameters (prothombin time/international normalized ratio, activated partial thromboplastin time, FVII clotting activity, platelet count, fibrinogen) | After 30 days
Presence of and/or de novo appearance of inhibiting antibodies to FVII | Prior to dosing
Presence of and/or de novo appearance of inhibiting antibodies to FVII | After 30 days
Number of Adverse Events | Until Day 5
Number of Serious Adverse Events | Until Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (16):
- Novo Nordisk Investigational Site, Princeton, New Jersey, United States
- Novo Nordisk Investigational Site, Paris La Défense Cedex, France
- Novo Nordisk Investigational Site, Mainz, Germany
- Novo Nordisk Investigational Site, Vouliagment, Greece
- Novo Nordisk Investigational Site, Kowloon, Hong Kong
- Novo Nordisk Investigational Site, Bangalore, India
- Novo Nordisk Investigational Site, Tehran, Iran
- Novo Nordisk Investigational Site, Kfar Saba, Israel
- Novo Nordisk Investigational Site, Rome, Italy
- Novo Nordisk Investigational Site, Karachi, Pakistan
- Novo Nordisk Investigational Site, Belgrade, Serbia
- Novo Nordisk Investigational Site, Bratislava, Slovakia
- Novo Nordisk Investigational Site, Madrid, Spain
- Novo Nordisk Investigational Site, Bangkok, Thailand
- Novo Nordisk Investigational Site, Istanbul, Turkey (Türkiye)
- Novo Nordisk Investigational Site, Caracas, Venezuela

REFERENCES:
- [Result] Mariani G, Dolce A, Batorova A, Auerswald G, Schved JF, Siragusa S, Napolitano M, Knudsen JB, Ingerslev J; STER and the International Factor VII Deficiency Study Groups. Recombinant, activated factor VII for surgery in factor VII deficiency: a prospective evaluation - the surgical STER. Br J Haematol. 2011 Feb;152(3):340-6. doi: 10.1111/j.1365-2141.2010.08287.x. Epub 2010 Dec 16. PMID 21158750
- [Result] Mariani G, Dolce A, Napolitano M, Ingerslev J, Giansily-Blaizot M, Di Minno MD, Auerswald G, De Saez AR, Tagliaferri A, Batorova A; STER (Seven Treatment Evaluation Registry). Invasive procedures and minor surgery in factor VII deficiency. Haemophilia. 2012 May;18(3):e63-5. doi: 10.1111/j.1365-2516.2012.02751.x. Epub 2012 Feb 22. No abstract available. PMID 22356641
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com